CLINICAL TRIAL: NCT06827795
Title: An Open, Parallel-group, Randomized, Medical Device Study to Assess the Usability and Performance of Surgify HaloTM in Spine Surgery Versus State-of-art (Rosen Burr)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Surgify Medical Oy (Industry)
Collaborators: North Shore University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00079896
Record Dates: First submitted 2025-01-09; First posted 2025-02-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Spine Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Surgify Halo (Other)
  Interventions: Device: A burr used in spine surgery
- State of art Rosen burr (Other)
  Interventions: Device: A burr used in spine surgery

INTERVENTIONS:
Device: A burr used in spine surgery — A burr used in spine surgery

SUMMARY:
The purpose of this research study is to:

test the usability and performance of the medical device Surgify Halo ™ in revision spine surgery test the level of "chattering " during the use of the device test the cutting performance of Surgify Halo™in comparison to the usual drill bit used in spine surgery ( Rosen burr).

This medical device is available for its indications for shaping and removal of hard tissue and bone in neurosurgical, spinal, ENT, and general surgical procedures.

The target is to enroll 30 participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Disease of the spine or head requiring surgery with bone removal

  * Ability to understand the purpose and risks of the study and to give written informed consent
  * Age 21-85 years

Exclusion Criteria:

* Previous surgery in the same area

  * Abnormalities of bone tissue
  * Vulnerable patients (such as prisoners, Individuals with limited or no reading skills, decisionally impaired persons, persons in nursing homes, patients in emergency), and pregnant women
  * Allergy or hypersensitivity to medical-grade stainless steel or any alloying components
  * Problems with blood clotting

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Usability and performance of the medical device Surgify Halo ™ in revision spine surgery | From enrollment to the end of the surgery until the end of the stay in the recovery room.
  Test the level of "chattering " during the use of the device and test the cutting performance of Surgify Halo™ in comparison to the usual drill bit used in spine surgery ( Rosen burr)

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided